## NCT04887129

## **October 1,2024**

## **DATA and STATISTICAL ANALYSIS**

Title: COV-IDD: Testing for COVID-19 in high risk children with intellectual and

developmental disabilities

**Principal Investigator:** 

John Foxe, PhD

**Department of Neuroscience** 

## **DATA and STATISTICAL ANALYSIS**

Primary data analysis will focus on understanding the spread of COVID-19 in a school for children with Intellectual and developmental Disabilities. By testing both students and staff in the school, and understanding interactions of staff and students throughout the day we aim to understand risk and develop risk mitigation techniques to help the school better reduce outbreaks and risk of infection. Based on blood samples we will also study the immune response of students and staff both to vaccination and also to infection. The time course of the immune response will be evaluated. Information about immune responses and infection will be conveyed to families and staff in order to encourage vaccination and also to help them understand how they may be putting their students and families at risk. Longitudinal and regular virological testing will track infection rates, and serological testing will quantify the durability of protective immunologic responses, which may be shorter-lived in IDD populations.

Statistical analyses will be performed using SPSS, or other similar software. Descriptive statistics will describe the incidence rates of COVID infection in participants, and the immunity levels of the students and staff (based on serological testing). Network modelling and agent-based simulations will be used to interactively test mitigation strategies. Qualitative surveys of participants will facilitate understanding of key community concerns, myths, and misconceptions about vaccination, with a goal of developing a multimodal educational campaign that addresses these concerns.